CLINICAL TRIAL: NCT06872411
Title: Evaluating Acceptability and Feasibility of an Enhanced Digital Intervention for Preventing Postpartum Mental Health Difficulties in Fathers
Brief Title: Evaluating a Mental Health Digital Intervention for Dads
Acronym: HealthyDads
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Deborah Da Costa, Deborah Da Costa, PhD, Associate Professor, Department of Medicine, McGill University; Scientist, RI-MUHC, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-11066
Record Dates: First submitted 2025-02-26; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HealthyDads web-based program group (Experimental): All participants in the study will be asked to use the HealthyDads website which includes up-to-date information and strategies related to i) prevention or reduction of stress and depressive symptoms; ii) parenting skills preparation tailored to expectant dads and iii) healthy lifestyle promotion for men at risk for depression.
  Interventions: Other: HealthyDads Digital Intervention

INTERVENTIONS:
Other: HealthyDads Digital Intervention — HealthyDads is a prototype bilingual self-guided psychoeducational Digital Intervention with accurate and easily accessible information on topics related to mental health, parenting and health behaviors, along with strategies to optimize each.

SUMMARY:
Approximately one in 10 fathers experience mental health difficulties during their partner's pregnancy and/or the postpartum period. There is a need for routine depression screening and timely interventions for fathers in the postpartum however there is a lack of resources tailored to men. To fill this gap, the investigators developed HealthyDads which includes up-to-date information and strategies related to i) prevention or reduction of stress and depressive symptoms; ii) parenting skills preparation tailored to expectant dads and iii) healthy lifestyle promotion for men at risk for depression. The investigators objective is to evaluate the acceptability of the HealthDads website targeting the mental health of at risk expectant fathers.

ELIGIBILITY:
Inclusion Criteria:

Fathers-to-be who:

* reside in Canada
* able to communicate in French or English
* gestational age of partner's pregnancy between 14-28 weeks
* internet access
* score <12 on the EPDS
* at least 1 risk factor for depression if they score <6 on the EPDS: a) history of depression; b) elevated anxiety (score >10 on the Generalized Anxiety Disorder 7-item (GAD-7) scale)116; or c) couple discord (established cutoff score <13 on the 4-item Dyadic Adjustment Scale117 or Pittsburgh Sleep Quality Index global score >5

Exclusion Criteria:

* suicidal ideation or intent
* score ≥12 on the EPDS
* having a severe psychiatric disorder as reported by the participant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Engagement with Digital Intervention: Number of Logins | From enrollment to the end of the intervention at 6 weeks
  To evaluate participant engagement with the digital intervention HealthDads, the investigators will track the number of times the participant logs into the intervention.
Intervention Acceptability and Expectancies Questionnaire (IAEQ) | From enrollement to the end of the intervention at 6 weeks
  Evaluates users' acceptance of the DI and potential barriers and facilitators to acceptance. Scale of minimum value 1 to a maximum value of 5 where a higher score indicates a better outcome.
Engagement with Digital Intervention: Number of modules viewed | From enrollment to the end of the intervention at 6 weeks
  In order to evaluate the engagement with the digital intervention HealthDads, the investigators will track the number of modules each participant views.
Engagement with Digital Intervention: Total number of pages viewed | From enrollment to the end of the intervention at 6 weeks
  In order to evaluate the engagement with the digital intervention HealthDads, the investigators will track the total number of intervention pages each participant views.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | From enrollment to the end of follow-up at 12 months following the birth of their baby
  The Edinburgh Postnatal Depressive Scale is a 10 question screening tool used to evaluate depressive symptoms. The minimum score is 0 and maximum is 30 with a higher score indicating more severe depression.
Male Depression Risk Scale (MDRS-22) | From enrollment to the end of follow-up at 12 months following the birth of their baby
  The Male Depression Risk Scale will assess masculine depressive symptoms. The minimum score is 0 and maximum is 154 with higher scores indicative of a greater risk of significant depressive symptoms.
Generalized Anxiety Disorder 7-item (GAD-7) | From enrollment to the end of follow-up 12 months after the birth of their baby
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is scored from 0 to 21, with higher scores indicating more severe anxiety.

IPD SHARING:
Plan to Share IPD: Undecided